CLINICAL TRIAL: NCT04939350
Title: Evaluation of the Vaccination Coverage in a Prospective Cohort of Cirrhotic Patients Followed in the General Hospitals in France in 2021 and in 2022.
Brief Title: Evaluation of the Vaccination Coverage of Cirrhotic Patients Followed in the General Hospitals in France in 2021
Acronym: VACCIR
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Sud Francilien (Other)
Responsible Party: Sponsor
Other Study IDs: IDRCB 2021-A00343-38
Record Dates: First submitted 2021-06-15; First posted 2021-06-25 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Cirrhosis
Keywords: Vaccinal coverage; vaccination; cirrhosis; cirrhotic; COVID; hepatitis B; hepatitis A; influenzae virus; pneumococcus; tetanus; poliomyelitis
MeSH Terms: conditions — Fibrosis; Hepatitis B; Hepatitis A; Tetanus; Poliomyelitis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionnaire — patients will complete a vaccination questionnaire

SUMMARY:
the purpose of this study is to estimate vacinal coverage against hepatitis A and B viruses, pneumococcus, diphtheria/tetanos and poliomyelitis, influenza virus and covid in cirrhotic patients followed in general hospitals of France and to show the

DETAILED DESCRIPTION:
Cirrhosis is a serious liver disease very common in France, affecting nearly 200,000 people. These patients have an impaired immune response. They are, therefore, more frequently prone to bacterial, viral and fungal infections and these are more severe with high mortality. 30-50% of cirrhotics admitted to a hospital ward have sepsis, with pneumococcal bacterial infections being particularly severe. The risk of developing seasonal influenza is 5.7 times higher in cirrhotics with a risk of mortality multiplied by 169. COVID19 infection is responsible for a very high mortality (34%) in case of severe resuscitation form. Acute infections with hepatitis A (HAV) and B (HBV) viruses frequently lead to worsening liver failure decompensating to cirrhosis, and sometimes life-threatening fulminant hepatitis. Finally, chronic infection with the hepatitis B virus combined with another etiology of cirrhosis accelerates the course of liver disease and promotes the occurrence of hepatocellular carcinoma.

Limiting the incidence of viral and bacterial infections in these patients is crucial. The High Authority of Health (HAS) published recommendations in 2007 advising patients with cirrhosis vaccinations against hepatitis A and B viruses, influenza and against bacterial pneumococcal infections, confirmed by the High Council of Public Health.

There are few data on vaccination coverage among cirrhotic patients. An unpublished French study from 2000 revealed low vaccination rates: 34% for pneumococcus, 55% for influenza, 32 to 42% for the hepatitis B virus and 20 to 38% for the hepatitis A virus. No recent studies have assessed the impact of the HAS recommendations.

The purpose of this study is to estimate vacinal coverage against hepatitis A and B viruses, pneumococcus, diphtheria/tetanos and poliomyelitis, influenza virus and covid in cirrhotic patients followed in general hospitals of France

ELIGIBILITY:
Inclusion Criteria:

* adult patient
* histologically proven or asserted cirrhosis on a combination of clinical, biological, endoscopic and radiological criteria
* follow-up of cirrhosis > 6 months
* subject informed of the study and not having objected to it.

Exclusion Criteria:

* immunosuppression not related to liver disease: HIV, variable common immune deficiency, chemotherapy, anatomical splenectomy, immunosuppressive treatments for non-hepatic disease
* vaccine contraindication.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All cirrhotic patients followed for at least 6 months in consultation or hospitalization during the duration of the study in the general hospitals members of the ANGH participating in the study.
Sampling Method: Probability Sample
Enrollment: 742 (Actual)
Dates: Start 2021-09-27 (Actual); Primary Completion 2022-12-27 (Actual); Study Completion 2022-12-27 (Actual)

PRIMARY OUTCOMES:
percentage fully immunization coverage | Day 0
  percentage of patients fully vaccinated against polio DT, seasonal influenza, HAV, HBV, pneumococcal and COVID19 in our sample

SECONDARY OUTCOMES:
percentage DTpolio immunization coverage | Day 0
  Percentage of vaccination against DTPolio
percentage HAV immunization coverage | Day 0
  Percentage of vaccination against HAV
percentage HBV immunization coverage | Day 0
  Percentages of vaccination against HBV
percentage Pneumococcal immunization coverage | Day 0
  Percentages of vaccination against pneumococcaL
percentage Influenza virus immunization coverage | Day 0
  Percentage of vaccination against seasonal influenza
percentage COVID immunization coverage | Day 0
  Percentage of vaccination against COVID19

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Sud Francilien, Corbeil-Essonnes, France

IPD SHARING:
Plan to Share IPD: No